CLINICAL TRIAL: NCT01782170
Title: Phase II Study: Evaluate Efficacy of Iocide Oral Rinse in a Human Clinical Trial of Gingival Inflammation and Investigate Effects on Biological Markers Indicative of Systemic Disease
Brief Title: Efficacy of Iocide Oral Rinse Against Gingival Inflammation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UK12-0972-F2L; R44HL101821 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Gingivitis; Investigation of Biological Markers of Inflammation
Keywords: Gingivitis; Biomarkers; Biological Markers of Inflammation
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iocide Oral Rinse (Active Comparator): Iocide Oral Rinse once daily 30 second rinse for 24 weeks
  Interventions: Drug: Iocide Oral Rinse
- Placebo Control (Placebo Comparator): Once daily 30 second rinse for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iocide Oral Rinse
  Other Names: Iocide Oral Rinse - once daily 30 second rinse for 24 weeks
  Arms: Iocide Oral Rinse
Drug: Placebo
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to explore the efficacy of Iocide oral rinse in a human clinical trial of gingivitis. Iocide oral rinse will be evaluated against a placebo rinse. Indices for gingivitis, plaque and bleeding will be scored and blood tests will be performed to determine the effect of the antimicrobial oral rinse on relative levels of biological markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

Subjects shall meet all of the following inclusion criteria to be eligible for participation in this study:

* Males or non-pregnant females of at least 18 years of age, and in good general health, as determined by Investigator;
* Have at least 16 natural, gradable teeth and good dental health, as determined by Investigator;
* Have > 25% sites with Gingival Index (GI) scores of > 2 at Visits 1 and 2;
* Have Plaque Index (PI) scores of > 1 on > 50% of sites;
* Use of effective method of contraception for the duration of the study or permanently sterilized;
* Able and willing to comply with study requirements including following instructions on study treatment and returning for follow-up visits as required by the protocol;
* Have full understanding of all elements of, and signature and dating of the written informed consent prior to the initiation of protocol specified procedures;
* Females with childbearing potential must have a negative pregnancy test before and during the study period. Sexually active females must be using an effective form of birth control or abstinence. These methods include oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrol implants (Norplant®), medroxyprogesterone acetate injections (Depo-provera®) or contraceptive foam with a condom.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be eligible for participation in this study:

* History, or current evidence, of any significant acute or chronic subject-reported medical or psychiatric condition that, in the opinion of the Investigator, would render examination difficult or invalid or prevent the subject from active study participation;
* ≤24% of sites with GI score >2;
* Thyroid peroxidase antibody (TPOab) positive >34;
* Screening serum level of thyroid stimulating hormone (TSH) <0.45 or >4.5;
* Treatment with antibiotic within the one (1) month period prior to the screening examination;
* History of heart murmur, history of rheumatic fever, valvular disease, prosthetic implant or any other condition requiring antibiotic premedication;
* History of thyroid disease;
* Purported sensitivity or allergy to iodine;
* Known sensitivity or allergy to shellfish;
* History of diabetes;
* History of autoimmune disease;
* Gross oral pathology (periodontal disease, rampant caries, tissue damage created by poor oral care or treatment, soft or hard tissue tumors) that, in the opinion of the Investigator, could influence the outcome of the study;
* True periodontal pockets of > 5 mm and/or visible recession indicative of attachment loss;
* Current signs or symptoms of mucosal tissue ulcerations or inflammation, or canker sores;
* Presence of orthodontic appliances or any removable appliance that impinges on the oral tissues being assessed;
* History of early onset periodontal disease or acute necrotizing ulcerative gingivitis;
* Subject reported history in past 6 months or current alcohol abuse that, in the opinion of the Investigator, could influence the outcome of the study;
* Subject reported history of last past 6 months or current drug abuse;
* Chronic treatment (2 weeks or more) with any medication known to affect periodontal status (including phenytoin, calcium antagonists, cyclosporine, coumarin, non-steroidal antiinflammatory drugs, and aspirin) within 1 month of the screening examination. All other medications for chronic medical conditions have been initiated at least 3 months before enrollment;
* Current use of a statin or the use of a statin within the past sixty (60) days of screening;
* Concomitant therapy with another investigational drug or device without prior approval from the Sponsor within four weeks prior to Visit 2 (Study Day 1);
* Concomitant endodontic or periodontal therapy other than prophylaxis in the past six (6) months;
* Females with childbearing potential with a positive pregnancy test, pregnant or nursing mothers, suspected pregnancy, or intention to become pregnant during the study;
* Residence in the same household as a subject already enrolled in the study (inclusion may create blinding and/or compliance issues);
* Unable and unwilling to comply with the informed consent process, to meet study requirements including following instructions on study intervention, and to return for follow-up visits as required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Gingival Index (GI) | Study Days -21 to -7 through Study Day 168

SECONDARY OUTCOMES:
Change in Biological Marker Data | Study Day 1, Day 28, Day 84 and Day 168

OTHER OUTCOMES:
Assessment of Product Safety | Study Days 1 through Study Days 168
  The assessment of product safety will include the following: incidence of adverse events, measures of thyroid function, and iodine excretion. Additionally, investigators will assess any development of opportunistic infection with Candida albicans, changes in oral tissues, and concomitant medication interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Dolphus R Dawson III, DMD, MS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Center for Oral Health Research, College of Dentistry, Lexington, Kentucky, United States